CLINICAL TRIAL: NCT00102674
Title: The Pharmacokinetics and Pharmacodynamics of a Cangrelor Bolus Plus Infusion in Healthy Volunteers
Brief Title: Pharmacokinetics/Pharmacodynamics (PK/PD) of Cangrelor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-CAN-04-02
Record Dates: First submitted 2005-01-31; First posted 2005-02-01 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2005-03

CONDITIONS: Healthy
Keywords: cangrelor; clopidogrel
MeSH Terms: interventions — cangrelor

INTERVENTIONS:
Drug: cangrelor

SUMMARY:
The purposes of this study are to:

* Evaluate the tolerability of two cangrelor regimens.
* Compare the PD of cangrelor regimens with oral clopidogrel.

DETAILED DESCRIPTION:
The purposes of this study are:

* To evaluate the tolerability of two cangrelor regimens of bolus plus infusion (A and B).
* To characterize the pharmacokinetics of Cangrelor (A and B).
* To compare the pharmacodynamics of cangrelor regimens with that of an oral 600 mg dose of clopidogrel (A, B, C and D).
* To determine the effect of prior cangrelor treatment on the pharmacodynamics of clopidogrel (C and D).
* To determine the effect of prior clopidogrel treatment on the pharmacodynamics of cangrelor (Group D).
* To determine the effects of concomitant clopidogrel and cangrelor exposure on the pharmacodynamics of clopidogrel (Group D).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent before initiation of any study related procedures.
* Age 18 - 55 years
* Normal findings on physical examination.
* A normal 12-lead ECG and normal vital signs (blood pressure, heart rate), unless any abnormality was considered clinically irrelevant by the investigator.
* Normal laboratory and hematology values unless the investigator considered an abnormality to be clinically irrelevant.
* Negative test for pregnancy as determined by urinary b-HCG prior to the administration of study drug for all females of child-bearing potential.
* Body Mass Index (BMI) between 20 and 25 kg/m2 based on actual body weight.

Exclusion Criteria:

* A history of or presence of renal, hepatic, neurological, hematological, gastrointestinal, or psychiatric disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Hypersensitivity to clopidogrel or cangrelor (or the excipients therein).
* Symptoms of a clinically significant illness, or surgery or trauma within 3 months prior to screening.
* Donation of blood or plasma totaling more than 500 mL within the 3 months preceeding the study.
* A significant history of alcohol or drug abuse, a positive urine drug screen, tobacco use within the 3 months preceding enrollment, or alcohol ingestion within 48 hours of dosing.
* A history of hepatitis or human immunodeficiency virus (HIV) or exposure thereto.
* Use of any prescribed medications in the 2 weeks prior to dosing, any aspirin or naproxen-containing medication within 2 weeks of dosing, use of acetaminophen within 24 hours or ibuprofen, vitamins or dietary supplements within 48 hours of dosing (oral contraceptives are permitted).
* Personal or family history of coagulation or bleeding disorders, or reasonable suspicion of vascular malformations, including aneurysms; history of important bleeding, (i.e. hematemesis, rectal bleeding, melena, severe or recurrent epistaxis, hemoptysis or intracranial hemorrhage), history of head injury or intracerebral disease, or recent or planned spinal or epidural puncture.
* Significant epigastric pain or "indigestion", either chronically or within 4 weeks prior to screening.
* Diagnosed hypertension, or supine blood pressure at or above 150/90 mmHG or less than 100/50 mmHg at screening.
* Participation in any clinical study with an investigational new drug in the 3 months prior to dosing in the study or participation in a study with a new formulation of a marketed drug in the previous 3 months.
* Anemia or thrombocytopenia (values on screening hematology less than the reporting laboratory's lower limit of normal).
* Any other characteristic or condition which, in the opinion of the investigator, makes participation in this study inappropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-03; Study Completion 2005-05

PRIMARY OUTCOMES:
To evaluate the tolerability of two cangrelor regimens

CONTACTS AND LOCATIONS:
Overall Officials: Steven Steinhubl, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States